# **Study protocol:**

Title of Project: Internet-based cognitive behaviour therapy for adults with tinnitus in the United Kingdom

**Trial registration**: ClinicalTrials.gov; NCT02370810, date 05/03/2015

Ethical approval: Research Ethics Committee (REC) of Anglia Ruskin University

(FST/FREP/14/478)

Author: Eldré W. Beukes,

Date: 17 September 2015

## **INTRODUCTION**

Tinnitus is one of the most distressing and debilitating hearing-related symptoms.<sup>1</sup> Unwanted sounds, such as ringing or buzzing are experienced, in the absence of a concurrent external sound source.<sup>2</sup> It is highly prevalent, affecting between 10-15% of adults in the UK, with an increased prevalence in older adults.<sup>3</sup>

Despite much research, medical treatments are usually ineffective at reducing tinnitus and a cure remains to be found. Tinnitus is therefore managed as a chronic condition, thereby adding strain on current healthcare systems. For some, experiencing tinnitus can result in a complex set of complaints. As there is a strong relationship between tinnitus and hearing difficulties, this adds to the distress experienced. In addition to the possible adverse effects on daily life, such as the impact on sleep, mood and concentration, there may also be a number of indirect psychological and psychosocial effects, including depression and anxiety. These concurrent physical and psychological effects add to the healthcare burden, as further input may be required from various health professionals.

When it comes to tinnitus management strategies, there is a low evidence-base for many practices. Of Good Practice Guidelines for tinnitus management were set by the Department of Health in the UK in 2009. Hoare and colleagues, found poor guideline adherence, unequal access to care, lack of standardization and limited use of psychological interventions for tinnitus. Innovative ways of addressing these issues in the UK are therefore required.

Cognitive Behavioural Therapy (CBT) is a technique, which reduces the distress associated with tinnitus, <sup>13</sup> and is one of the tinnitus treatment options with the most evidence of effectiveness. <sup>14</sup> It has been shown to add to the efficacy of Audiology/ENT approaches to treatment. <sup>15</sup> It is however, rarely offered in clinical practice, <sup>16</sup> particularly in the UK. <sup>17</sup> This is largely due to a shortage of those with appropriate CBT training, such as Psychologists who are audiologically literate, and willing to manage tinnitus. <sup>18</sup>

To provide an accessible evidence-based tinnitus treatment, an internet-based, CBT intervention (iCBT) was developed by Andersson and colleagues, <sup>19</sup> and results of their initial Randomized Control Trial (RCT) showed promising effects. Following intervention improvements, further studies, run in Sweden and Germany, indicated similar results to face-

to-face group CBT.<sup>20,21</sup> A further RCT in Australia by Abbott and colleagues,<sup>22</sup> found results of iCBT did not show any statistically significant benefit over a information-only control program (without CBT content). In addition, the attrition rate was higher in the iCBT group. This poses questions regarding whether the structure and presentation of the intervention requires updating to improve overall outcomes. If iCBT for tinnitus distress was feasible in the UK it may bridge a gap for those who have not been able to access appropriate tinnitus services. It could furthermore reduce the burden on the healthcare system for those who do not require supra-specialist support.

A study to determine whether iCBT could be a suitable intervention is therefore of value. The aim of this study is to further our knowledge of the feasibility and effectiveness of iCBT for tinnitus management in the UK. This research is timely and in line with two of the tinnitus research priorities recommended by the James Lind Alliance,<sup>4</sup> namely: research investigating which management strategies are more effective than the usual model of audiological care in improving outcomes for people with tinnitus and research determining whether CBT, delivered by audiology professionals, is effective for people with tinnitus.

The research objectives for this study are therefore as follows:

- 1. To establish the feasibility of using iCBT for tinnitus distress, as an intervention for adults with tinnitus in the UK
- 2. To evaluate the effectiveness of iCBT for tinnitus distress in reducing the impact associated with tinnitus for adults in the UK.
- 3. To ascertain predictors of outcome for whom this iCBT intervention is a suitable intervention
- 4. To determine the longer term effects of iCBT, 12 months post-intervention

## **METHODS**

## Study design

This will be an internet-based study run in the UK. This intervention study will be implemented as a two-armed RCT, with a one-year follow-up, to evaluate the effectiveness iCBT on tinnitus distress. An effectiveness trial has been selected, to increase the extent to which the study results can be generalised and be used to identify for which subgroups of tinnitus sufferers this is a suitable intervention. A delayed treatment design using a weekly check-in control (WCI) group will be used, as shown in Figure 1. The objective is to test the superiority of the

intervention, with the hypothesis that the treatment group will perform better than the weekly check-in group. These groups will be followed prospectively for 1 year, to establish the long-term effectiveness of the intervention programme.

This study design is described using the Standard Protocol Items, Recommendations for Interventional Trials (SPIRIT) checklist.<sup>23,24</sup> and has been registered with Clinical Trials.gov: NCT02370810, date 05/03/2015



# Study groups

There will be two study groups. The *Test Group* will receive the eight-week long iCBT treatment following baseline measurements and allocation (after  $T_0$ ). The weekly check-in *Control Group* will be monitored during the active treatment phase by means of the Tinnitus

Handicap Inventory- Screening Version.<sup>25</sup> but will have no other contact or involvement in the study during this period. The control group will undergo the same iCBT intervention once the treatment group finishes the programme (after T<sub>1</sub>).

### **Inclusion Criteria**

A clinical evaluation prior to partaking in the study is desirable, to rule out the presence of a serious auditory pathology or associated psychological problem, which may be related to having tinnitus.<sup>26</sup> If there are any concerns, a letter will be provided for participants to take to their General Practitioner, for further management.

Participant's eligibility for the study is as follows:

- i) Aged 18 years and over living in the UK
- ii) The ability to read and type in English
- No barriers to using a computer (e.g. significant fine motor control or visual problems)
- iv) Internet and e-mail access, and the ability to use these
- v) Commitment to completing the programme
- vi) Completion of the online screening and outcome questionnaires
- vii) Agreeing to participate in either group and be randomized to one of these groups
- viii) Understanding and working towards the end goal of reducing the impact and distress of tinnitus, although the strength of the tinnitus may remain the same
- ix) Be available for 12 months after starting the study to complete a 1 year follow-up questionnaire
- x) Suffering with tinnitus for a minimum period of 3 months
- xi) Tinnitus outcome measure scores indicating the need for tinnitus care (26 or above on the Tinnitus Functional Index)<sup>27</sup>

## **Exclusion Criteria**

- i) Reporting any major medical or psychiatric conditions
- ii) Reporting pulsatile, objective or unilateral tinnitus, which have not been investigated medically
- iii) Tinnitus as a consequence of a medical disorder, still under investigation
- iv) Undergoing any tinnitus therapy concurrently to partaking in this study

A two-staged selection procedure will be followed:

- i) An online screening questionnaire, which includes health and mental health related questions
- ii) A telephone interview, during which the researcher will re-check eligibility and provide the opportunity for potential participants to ask any questions related to the study.

## Recruitment

Recruitment will be UK wide, using as many different forms as possible to achieve adequate participant enrolment. Information about the study will be advertised at tinnitus and hearing-related support groups and charities, in their newsletters and drop in centres. It will furthermore be advertised in Audiology Departments and by using social media. Talks to professionals, such as ENT Consultants and Audiologists, will also be given to introduce the study and aid recruitment. Those interested can obtain information and register interest on the study website.

# Sample size

Sample size estimation was calculated using Power and Sample Size Programme, version 3.1.2 and based on achieving a clinically relevant change of 13 points (std dev 24.7) in the main outcome measure to be used for this study; the Tinnitus Functional Index.<sup>27</sup> This indicated 30 participants were required per group; with an allocation ratio of 1:1, to achieve a two-sided significance level of 0.05 and effect size of 0.8. As these calculations are based on a fairly new outcome measure and there may be dropouts, an additional 40 participants will be added, to ensure enough valid data to draw conclusions from. Therefore, 70 participants will be assigned to the experimental group, and 70 participants to the control group. This is roughly in line with the sample sizes used in similar studies.

### Allocation

Participants will be randomly assigned to either control or experimental group with a 1:1 allocation using a computer generated randomization schedule (<a href="http://www.randomizer.org/">http://www.randomizer.org/</a>) by an independent researcher. To prevent an unequal distribution among groups, participants will be pre-stratified on the factors of age (<= 60 or >60 year) and Tinnitus severity (TFI <= 50 or >50). Furthermore, block randomization, with blocks of four, will be applied to ensure equal groups sizes within each stratum.

Following allocation participants will be contacted by telephone, to provide the opportunity to discuss the aspects of the study and answer any questions. This initial contact has been found to be valuable to ensure participants are motivated to complete the treatment.<sup>20</sup>

## Intervention

The intervention to be followed, is built on an internet-based CBT self-help programme (iCBT) for reducing tinnitus distress developed by Andersson and colleagues.<sup>19</sup> It incorporates a combination of a cognitive rational,<sup>28</sup> and a learning theory approach.<sup>29</sup> The original intervention was largely text based. The present authors have redesigned and modified the intervention content and presentation, to have an interactive e-learning version, as shown in Figure 2. This will ensure the intervention is visually stimulating, engaging and responsive to participant's progress.

The intervention consists of fixed and optional modules, covered over a period of 8 weeks, as shown in Table 1. The modules contain a mixture of information, videos, quizzes, diagrams, suggested techniques to apply to daily life, worksheets to keep track of progress, solutions for common problems and downloadable information.

The iCBT intervention will be delivered on a secure web platform, for which participants will receive password protected login information.

**Table 1: The components of the iCBT intervention** 

| Week | Module | Explanation | Application |
|---|---|---|---|
| 1 | About this treatment | Introduction to the modules | Reading |
| | Tinnitus overview | In depth information | Quizzes |
| 2 | Relaxation: step 1 | Deep relaxation | 10-15 min, twice/day |
| | Identifying negative | The link between thoughts and | Writing down thoughts |
| | thoughts | feelings | |
| | *Sound enrichment | Using background sounds | Applying external sounds |
| 3 | Relaxation: step 2 | Diaphragmatic breathing | 5-7 min, twice/day |
| | Cognitive restructuring | Analysing thoughts | Writing down situation, |
| | | | thoughts, feelings |
| | *Sleep guidelines | Various Techniques | Chose and apply |
| | | | techniques |

| 4 | Relaxation: step 3 | Entire body relaxation | 2-3 min, twice/day |
|---|---|---|---|
| | Positive imagery | Use to enhance relaxation | Twice/day after relaxation |
| | *Concentration tips | Techniques discussed | Engage in mentally |
| | | | engaging activities |
| 5 | Relaxation: step 4 | Rapid relaxation | 20-60 sec, 5-10 times/day |
| | Focus exercises | Mindful awareness | Twice/day after relaxation |
| | *Sensitivity to sound | Gradual exposure | Listen to non-damaging, |
| | | | non-annoying sounds |
| 6 | Relaxation: step 5 | Rapid relaxation in more | 30-60 sec, 10-15 times/day |
| | | difficult situations | |
| | Reinterpretation of | Change negative tinnitus | Writing about tinnitus |
| | tinnitus | associations | thoughts |
| | * Hearing tactics | Communication advice | Follow advice |
| 7 | Relaxation: step 6 | Making relaxation part of daily | Rapid relaxation 10-20 |
| | | routines and habits | times/day |
| | Exposure to tinnitus | Decrease negative emotions and | Actively listen to tinnitus |
| | | for 5-10 min, once/day, | |
| | | | after relaxation |
| 8 | Key points summary | Highlighting key concepts | Online quiz |
| | Future planning | Maintenance and relapse | Making a plan to use tools |
| | | prevention | in daily life |

Optional modules are marked with an \*

# **Monitoring progress**

Participants will be minimally guided via a secure online messaging system. This therapeutic alliance will allow for feedback and assistance if participants have any difficulties and has shown better outcomes than internet interventions without this communication.<sup>30</sup> The clinician will contact any participants who have not completed their weekly progress worksheets to ensure they are assisted as required. In these worksheets, participants record details about when, where, and for how long they practiced the suggested techniques and how effective these techniques were.

As tinnitus therapy is largely delivered by the audiology community in the UK, an experienced Audiological Scientist, registered with the Health Professions Council, will therefore undertake the role of supporting the participants, to maintain consistency with the standard approach. Support will however be provided by a Psychologist, with experience in iCBT interventions and a protocol for dealing with different situations will be used.

### Assessment

The assessment battery will consist of a screening eligibility questionnaire and relevant self-reported outcome measures, related to areas which may be affected by tinnitus. Outcome measures for tinnitus severity, hearing handicap, insomnia, cognitive functioning, hyperacusis, anxiety, depression and life satisfaction were therefore selected. Careful consideration was given to ensure each questionnaire was as brief as possible and had good psychometric properties as seen in Table 2. The outcomes were furthermore selected to be aligned with the International Classification of Functioning, Disability and Health (ICF)<sup>31</sup> framework on the domains of activity limitation and participation restriction.

# The assessment battery and outcome measures will include:

- Eligibility screening: A range of demographic, tinnitus specific and health related
  questions will be asked to determine demographic variability and study eligibility.

  Open-ended questions asking about positive and negative experiences related to
  having tinnitus will also be incorporated.
- 2. The main outcome measures: The Tinnitus Functional Index (TFI), has been selected to determine tinnitus severity, as it is validated for assessing responsiveness to treatment both for scaling the severity and negative impact of tinnitus and for measuring treatment-related changes in tinnitus.<sup>27</sup> The TFI was specifically designed to measure the effectiveness of interventions, a feature lacking in previous tinnitus outcome measures.<sup>32</sup> Due to its validation for assessing treatment responsiveness, it was chosen above some other more established questionnaires, such as the Tinnitus Handicap Inventory.<sup>33</sup>

## 3. Secondary outcome measures:

3.1 The Tinnitus Handicap Inventory -Screening Version (THI-S),<sup>25</sup> will be used as a concise outcome measure, particularly to monitor tinnitus handicap on a weekly basis during the active treatment phase.

- 3.2 As there is a strong relationship between tinnitus and hearing difficulties,<sup>7</sup> the Hearing Handicap Inventory for Adults-Screening Version (HHIA-S),<sup>34</sup> will be administered to quantify perceived hearing handicap. It includes both emotional and social/situational subscales.
- 3.3 As sleep disturbances are commonly associated with tinnitus,<sup>35</sup> the Insomnia Severity Index (ISI)<sup>36</sup> will be included. This questionnaire assesses the nature, severity, and impact of insomnia by assessing sleep duration, sleep quality, the negative impact on daily functioning and psychological well-being.
- 3.4 As having tinnitus may disrupt cognitive functioning,<sup>37</sup> the Cognitive Failures questionnaire (CFQ)<sup>38</sup> will be included. It was designed to assess proneness to committing cognitive slips and errors in the completion of everyday tasks such as failures in perception, memory, and motor function.
- 3.5 As there is a high comorbidity of hyperacusis (a reduced tolerance of everyday sounds)<sup>39</sup> in those with tinnitus,<sup>40</sup> the Hyperacusis Questionnaire<sup>41</sup> will be administered. Although further work on the structure of this questionnaire is required to establish its reliability for measuring hyperacusis in the tinnitus research population, the scores obtained will be useful to compare pre and post-intervention changes.
- 3.6 As anxiety and depression are common comorbid conditions in individuals with tinnitus,<sup>6</sup> the Patient Health Questionnaire (PHQ-9),<sup>42</sup> to measure depression severity and the Generalised Anxiety Disorder (GAD-7),<sup>43</sup> to assess anxiety severity will be administered.
- 3.7 To include a measure of quality of life, the Satisfaction with Life Scales,<sup>44</sup> assessing global life satisfaction will be used. For the purpose of this study, it was felt that the questions in this scale were more appropriate than those of longer quality of life measures, which include areas of mobility and self-care, which are not directly targeted by this study.

Permission has been obtained to use the questionnaires, for which it is required, such as the TFI.

Table 2: Known psychometric properties of the questionnaires to be administered at some point during the study

| Measure and validation reference | Items | Scale used | Internal |
|---|---|---|---|
| | | | consistency |
| | | | (Cronbach's alpha) |
| Tinnitus Functional Index <sup>27</sup> | 25 | 1-10 | 0.97 |
| Tinnitus Handicap Inventory-Screening <sup>25</sup> | 10 | 1-3 | 0.87 |
| Hearing Handicap Inventory: Screening <sup>34</sup> | 10 | 1-3 | 0.93 |
| <b>Insomnia Severity Index</b> <sup>36</sup> | 7 | 0-4 | 0.74 |
| Cognitive Failures Questionnaire <sup>38</sup> | 25 | 0-4 | 0.89 |
| Hyperacusis Questionnaire <sup>41</sup> | 14 | 0-4 | 0.66-0.68 |
| Patient Health Questionnaire <sup>42</sup> | 9 | 0-3 | 0.83 |
| Generalised Anxiety Disorder <sup>45</sup> | 7 | 0-3 | 0.89 |
| Satisfaction with Life Scales <sup>44</sup> | 5 | 1-7 | 0.87 |

# **Questionnaire delivery**

The format of the questionnaire delivery will remain consistent throughout the study using online questionnaires. Not all questionnaires to be used have been validated for internet use. Previous research has found comparable results in terms of psychometric properties between computer and paper questionnaire delivery, with high test-retest reliability and completion rate on the internet. 46,47 See Table 3 for the schedule of outcome measure delivery.

## **Process Evaluation**

An intervention, such as iCBT is known as a 'complex intervention' as it combines different components but does not involve drugs or surgical procedures. To fully investigate the different aspects of this complex intervention, we will be exploring the processes involved in implementing the iCBT intervention, as shown in Figure 3, in parallel to the iCBT study. By integrating this process evaluation information with the outcome data, we will maximise our ability to interpret the results and the effectiveness of the intervention. 49

We will be combining components from three evaluation models, namely the Reach, Efficacy, Adoption, Implementation and Maintenance (RE-AIM model);<sup>50,51</sup> and those of Linnan and Steckler,<sup>52</sup> as well as those of Baranowski and Stables.<sup>53</sup> The following eight components have been selected:

- 1. *Recruitment:* procedures used to approach and attract participants.
- 2. *Reach:* the extent to which the targeted population were drawn to the study and were willing to be involved in this intervention study.

- 3. *Context:* characteristics of the participants that affect the iCBT intervention including social, demographical, socio-economic factors.
- 4. *Dose delivered:* The number of modules and component included in this iCBT intervention.
- 5. *Dose received:* The extent to which participants actively engage and interact with the resources provided by this iCBT intervention.
- 6. *Effectiveness:* examining both the positive and negative consequences of the intervention, as well as factors that may positively or negatively influence the effectiveness of the intervention from the participant's perspective.
- 7. *Maintenance*: keeping participants involved in this iCBT intervention and data collection.
- 8. *Fidelity*: The extent to which the intervention was implemented as planned.

These processes will be monitored during the intervention, by reflecting on study procedures and participant's experiences. After undergoing the intervention, participant satisfaction will be established using a Likert scale and telephone interview.

# Pilot study

All materials will be piloted prior to running the study. Both professionals and those with tinnitus will test all aspects of the platform. Likert scaled questionnaire will be administered, asking specific questions related to the suitability, usability, content and experiences with the intervention and questionnaires, together with open-ended questions. The aim will be to identify any hindrances regarding use of the platform and possible barriers to participation. If any major changes are required, the ethical committee and trial body will be notified.

Further feasibility measures will include the recruitment rates, retention of participants, compliance and acceptability of the intervention by participants. The feasibility of having an Audiological professional running the intervention under supervision, instead of a Psychologist will also be evaluated.

### **Data collection**

All data will be collected online. Baseline data will be collected at pre-treatment (- $T_1$ ), prior to allocation. During the active phase of the intervention, the 10 questions on the THI-S<sup>25</sup> will be collected on a weekly basis. Data will then be collected at post-treatment ( $T_1$ ) and after the control group completes the intervention ( $T_2$ ). To determine long-term effectiveness of the intervention, data will again be collected 12 months ( $T_x$ ) after the start of the intervention at close out, and this will end the study. The specific outcome measures for each collection point are shown in Table 3.

To improve attrition rates at follow-up, an e-mail will be sent to encourage participants to complete the questionnaires, with a maximum of three reminders. If they do not wish to further participate in the study, the reasons for their withdrawal will be recorded, where provided, by means of a post-treatment satisfaction questionnaire.

Table 3: Schedule of enrolment, interventions and assessment

| STUDY PERIOD | | | | | |
|---|---|---|---|---|---|
| | Enrolment | Allocation | Post-allocation | | Close-out |
| TIMEPOINT | -T <sub>1</sub> | $T_{\theta}$ | T <sub>1</sub> (8 weeks) | T <sub>2</sub> (16 weeks) | $T_x$ (1 year) |
| ENROLMENT | | | | | |
| Eligibility screen | X | | | | |
| Informed consent | X | | | | |
| Allocation | | X | | | |
| INTERVENTIONS | | | | | |
| Experimental group | | + | <b>—</b> | | |
| Control group | | | <b>—</b> | <b>—</b> | |
| ASSESSMENTS | | | | | |
| Tinnitus Functional Index | X | | X | X | X |
| Tinnitus Handicap Inventory-<br>Screening Version | X | X<br>(weekly) | X | X | X |
| Hearing Handicap Inventory-<br>Screening Version | X | | X | X | X |
| Insomnia Severity Index | X | | X | X | X |
| Cognitive Failures Questionnaire | X | | X | X | X |
| Hyperacusis Questionnaire | X | | X | X | X |

| Patient Health Questionnaire | X | X | X | X |
|------------------------------|---|---|---|---|
| Generalised Anxiety Disorder | X | X | X | X |
| Satisfaction with Life | X | X | X | X |

# **Data Management**

All participants will receive a non-traceable unique reference code to keep their identities blinded during the result analysis. All files used will be password protected. The researchers, statisticians and internal data monitoring committee (DMC), will have access to the final dataset. The DMC includes researchers who are independent to this study without competing interests. They will ensure accurate analysis and result interpretation.

# **Data Analysis**

Data analysis will be in accordance with Consolidated Standards of Reporting Trials (CONSORT) guidelines for randomized clinical trials.<sup>54</sup> The Statistical Package for Social Sciences (SPSS) version 20.0 will be used and the data analyst will be blinded to the groups, to minimise bias. Results at post-treatment will be based on an intention-to-treat paradigm, in which incomplete data sets will be analysed using multiple imputation, offered by SPSS. For all analyses, a two-tailed significance level of < 0.05 will be considered statistically significant. The data will be analysed, using a general linear model repeated measures approach to look at the effects of the intervention and changes over time.

Qualitative content analysis with a positivist philosophical approach will be used to analyse the responses for open-ended questions.<sup>55</sup> Integrating different analysis methods will yield further insight into the study outcomes.<sup>56</sup>

The study results will be shared in peer reviewed publications by the present authors and presented at research conferences. A summary of the findings will be available to study participants, members of tinnitus support and tinnitus charity groups.

## **Ethical considerations**

Ethical approval has been granted by the Research Ethics Committee (REC) of Anglia Ruskin University (FST/FREP/14/478). Participation is voluntary and all participants will provide

informed consent online. A full explanation of every step of the study and will given and participants will be able to withdraw at any stage without penalty.

A protocol has been established to ensure the security of participant's confidentiality on the web-portal, complying with European guidelines for internet studies. Participant's data will be anonymised as unique reference codes will be used. Protocols to minimise the risks to participants and the researcher have been put in place. The data, together with any other spontaneously reported adverse events during the intervention will be reported. If any participants were identified as requiring additional support, a letter will be provided for them to take to their General Practitioner, so that this care can be arranged.

## **DISCUSSION**

In this paper, the design of a study, to investigate the effectiveness and feasibility of an internet-based intervention for tinnitus in the UK, is outlined. The strength of the proposed methodology is the randomised design. A further strength is that not only the effects of the iCBT intervention, but also the process evaluation will be investigated, to fully determine the interventions feasibility and effectiveness.

This particular tinnitus intervention has been selected due to the numerous potential benefits it may have. It is a standardised treatment, in which each participant has access to the same materials. The researchers have however carefully considered how to improve on methods used in similar previous studies and built on these. The following improvements will be made during this study. Firstly, redesigning the module content and combining both CBT and audiology principles, thereby ensuring it is multidisciplinary in nature. Secondly, transforming the presentation of materials into an interactive e-learning version, which is visually stimulating may improve participant engagement. Thirdly, using a main outcome measure that is specifically designed for measuring intervention effects. Fourthly, assessing a range of outcomes to help identify for whom this intervention is most suited. Fifthly, enabling the intervention to be presented by an Audiologist instead of a Psychologist. Lastly, aiming for good participant retention by careful inclusion criteria and screening methods.

There are however potential barriers that can be forecasted for this study. Although according to the 2015 report from the Office of Statistics,<sup>57</sup> 86% of the population in Great Britain have

internet access, there is still a proportion who don't have access and will therefore not be able

to partake in this study. Those without access may be older adults, which might impact the

sample selected. There are also people with visual or motor disabilities who will be unable to

use a computer effectively, and therefore may not be suitable for this intervention unless they

have assistance. A further barrier is that participants will require motivation to complete the

questionnaires and treatment modules. A limitation of the study design is that it is not possible

to blind the researcher and participants during the intervention, as they will know in which

group they have been placed. Bias will however be minimized by stratification and blinding

during randomisation, and data analysis.

Feasibility and uptake of such an intervention will be determined by this study. It is however

encouraging that other internet based studies, run within the UK, for other health related

concerns, <sup>58,59</sup> have reported sufficient interest. Due to the multidisciplinary nature of the study,

it furthermore has the prospect of determining the effects of the iCBT intervention not only on

tinnitus outcomes, but also on the person globally, as various comorbid factors are being

investigated.

The potential impact of this research is that it can change the way in which tinnitus services

are delivered in the UK. If effective, iCBT may be suggested for certain tinnitus sufferers

following their clinical examination. This will address differential clinical demands and reduce

the number of tinnitus suffers needing face-to-face consultations. This may in turn diminish

the current burden on the NHS healthcare and lead to a significant potential cost saving to the

health service. It may also make treatment available to many who are unable to access speciality

tinnitus services

If this intervention is feasible, future studies should focus on comparing iCBT to the usual

tinnitus care in the UK. It is expected that the results of this study will become available early

in 2017.

Figure legends

Figure 1: Flow chart of the study design

Figure 2: The modified iCBT intervention

Figure 3: The processes to be evaluated following the study

17

### **Abbreviations**

**CBT-** Cognitive Behavioural Therapy

CFQ- Cognitive Failures Questionnaire

CONSORT- CONsolidated Standards of Reporting Trials

CSQ-8 - Client satisfaction questionnaire

DMC- data monitoring committee

DOH- Department of Health

GAD-7- Generalized anxiety Disorder

HFDTT- High Frequency Digit Triplet Test

HHIA-S – Hearing Handicap Inventory for Adults- Screening Version

**HQ-** Hyperacusis Questionnaire

iCBT- Internet based Cognitive Behavioural Therapy Intervention

ICF- International Classification of Functioning

ISI- Insomnia Severity Index

NHS- National Health System

PHQ-9 Patient Health Questionnaire

**REC-Research Ethics Committee** 

**RCT-Randomized Control Trial** 

SPIRIT-Standard Protocol Items, Recommendations for Interventional Trials

SPSS - Statistical Package for Social Sciences

SWLS- Satisfaction with Life Scales

TFI- Tinnitus Functional Index

THI-S- Tinnitus Handicap Inventory-Screening Version

UK – United Kingdom

WCI- weekly check-in control group

## **Funding**

This research received no specific grant from any funding agency in the public, commercial or not-for-profit sectors.

#### References

- 1. Cima RFF, Vlaeyen JWS, Maes IHL, Joore MA, Anteunis LJC. Tinnitus interferes with daily life activities: a psychometric examination of the Tinnitus Disability Index. Ear Hear 2011;32(5):623.
- 2. McFadden D. Tinnitus: Facts, theories, and treatments. : National Academies; 1982.
- 3. Davis A, Rafaie EA. Epidemiology of tinnitus. Tinnitus handbook 2000:1-23.
- 4. Hall DA, Mohamad N, Firkins L, Fenton M, Stockdale D. Identifying and prioritizing unmet research questions for people with tinnitus: the James Lind Alliance Tinnitus Priority Setting Partnership. Clin Invest 2013;3(1):21-28.

- 5. Maes IH, Cima RF, Vlaeyen JW, Anteunis LJ, Joore MA. Tinnitus: a cost study. Ear Hear 2013 Jul-Aug;34(4):508-514.
- 6. Belli S, Belli H, Bahcebasi T, Ozcetin A, Alpay E, Ertem U. Assessment of psychopathological aspects and psychiatric comorbidities in patients affected by tinnitus. European archives of oto-rhino-laryngology 2008;265(3):279-285.
- 7. Palmer KT, Griffin MJ, Syddall HE, Davis A, Pannett B, Coggon D. Occupational exposure to noise and the attributable burden of hearing difficulties in Great Britain. Occupational and environmental medicine 2002;59(9):634-639.
- 8. Bartels H, Middel BL, van der Laan BF, Staal MJ, Albers FW. The additive effect of co-occurring anxiety and depression on health status, quality of life and coping strategies in help-seeking tinnitus sufferers. Ear Hear 2008 Dec;29(6):947-956.
- 9. Cima RMJ, Joore M, Maes I, Scheyen D, Refaie E, Baguley DM, et al. Cost- effectiveness of multidisciplinary management of Tinnitus at a specialized Tinnitus centre. BMC Health Services Research 2009;9(1):29.
- 10. Hoare DJ, Kowalkowski VL, Kang S, Hall DA. Systematic review and meta-analyses of randomized controlled trials examining tinnitus management. Laryngoscope 2011;121(7):1555-1564.
- 11. Department of Health. Provision of services for adults with tinnitus. A good practice guide. London, England: Central Office of Information 2009.
- 12. Hoare DJ, Gander PE, Collins L, Smith S, Hall DA. Management of tinnitus in English NHS Audiology Departments: an evaluation of current practice. J Eval Clin Pract 2012;18(2):326-334.
- 13. Cima RF, Andersson G, Schmidt CJ, Henry JA. Cognitive-Behavioral Treatments for Tinnitus: A Review of the Literature. J Am Acad Audiol 2014;25(1):29-61.
- 14. Hesser H, Weise C, Westin VZ, Andersson G. A systematic review and meta-analysis of randomized controlled trials of cognitive—behavioral therapy for tinnitus distress. Clin Psychol Rev 2011;31(4):545-553.
- 15. Cima RF, Maes IH, Joore MA, Scheyen DJ, El Refaie A, Baguley DM, et al. Specialised treatment based on cognitive behaviour therapy versus usual care for tinnitus: a randomised controlled trial. The Lancet 2012;379(9830):1951-1959.
- 16. Gander PE, Hoare DJ, Collins L, Smith S, Hall DA. Tinnitus referral pathways within the National Health Service in England: a survey of their perceived effectiveness among audiology staff. BMC Health Serv Res 2011 Jul 6;11:162-6963-11-162.
- 17. Baguley D, McFerran D, Hall D. Tinnitus. The Lancet 2013;382(9904):1600-1607.
- 18. McFerran, D, Baguley, D. Is psychology really the best treatment for tinnitus? Clin Otolaryngoly 2009;34: 99–101

- 19. Andersson G, Strömgren T, Ström L, Lyttkens L. Randomized controlled trial of internet-based cognitive behavior therapy for distress associated with tinnitus. Psychosom Med 2002;64(5):810-816.
- 20. Jasper K, Weise C, Conrad I, Andersson G, Hiller W, Kleinstaeuber M. Internet-based guided self-help versus group cognitive behavioral therapy for chronic tinnitus: a randomized controlled trial. Psychother Psychosom 2014;83(4):234-246.
- 21. Kaldo V, Levin S, Widarsson J, Buhrman M, Larsen H-, Andersson G. Internet Versus Group Cognitive-Behavioral Treatment of Distress Associated With Tinnitus: A Randomized Controlled Trial. Behavior Therapy 2008;39(4):348-359.
- 22. Abbott JM, Kaldo V, Klein B, Austin D, Hamilton C, Piterman L, et al. A cluster randomised trial of an internet-based intervention program for tinnitus distress in an industrial setting. Cognitive behaviour therapy 2009;38(3):162-173.
- 23. Chan A, Tetzlaff JM, Altman DG, Laupacis A, Gøtzsche PC, Krleža-Jerić K, et al. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med 2013;158(3):200-207.
- 24. Chan A, Tetzlaff JM, Gøtzsche P,C., Altman DG, Mann H, Berlin JA, et al. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ: British Medical Journal 2013;346.
- 25. Newman CW, Sandridge, SA, Bolek L. Development and psychometric adequacy of the screening version of the tinnitus handicap inventory. Otol Neurotol. 2008; 29(3):276-81.
- 26. Baguley, D., Andersson, G., McFerran, D., & McKenna, L. "Medical Models of Tinnitus." *Tinnitus: A Multidisciplinary Approach, Second Edition*: 2012: 43-66. John Wiley & Sons.
- 27. Meikle MB, Henry JA, Griest SE, Stewart BJ, Abrams HB, McArdle R, et al. The tinnitus functional index: development of a new clinical measure for chronic, intrusive tinnitus. Ear Hear 2012 Mar-Apr;33(2):153-176.
- 28. Henry JL, Wilson PH. The psychological management of chronic tinnitus: a cognitive-behavioral approach. : Allyn & Bacon; 2001.
- 29. Hallam R, Rachman S, Hinchcliffe R. Psychological aspects of tinnitus. Contributions to medical psychology 1984;3:31-53.
- 30. Andersson G, Carlbring P, Berger T, Almlöv J, Cuijpers P. What makes internet therapy work? Cognitive Behaviour Therapy 2009;38(S1):55-60.
- 31. World Health Organization. International classification of functioning, disability and health. ICF GEnova, WHO 2001.
- 32. Kamalski DM, Hoekstra CE, van Zanten BG, Grolman W, Rovers MM. Measuring disease-specific health-related quality of life to evaluate treatment outcomes in tinnitus patients: A systematic review. Otolaryngology-Head and Neck Surgery 2010;143(2):181-185.

- 33. Newman CW, Jacobson GP, Spitzer JB. Development of the tinnitus handicap inventory. Archives of Otolaryngology–Head & Neck Surgery 1996;122(2):143-148.
- 34. Newman CW, Weinstein, BE, Jacobson, GP, Hug, GA. Test-retest reliability of the hearing handicap inventory for adults. *Ear and hearing*, 1991;12(5), 355-357.
- 35. Crönlein T, Langguth B, Geisler P, Hajak G. Tinnitus and insomnia. Prog Brain Res 2007;166:227-233.
- 36. Bastien CH, Vallières A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med 2001;2(4):297-307.
- 37. Andersson G, McKenna L. The role of cognition in tinnitus. Acta Otolaryngol 2006;126(S556):39-43.
- 38. Broadbent DE, Cooper PF, FitzGerald P, Parkes KR. The cognitive failures questionnaire (CFQ) and its correlates. British Journal of Clinical Psychology 1982;21(1):1-16.
- 39. Vernon JA. Pathophysiology of tinnitus: a special case--hyperacusis and a proposed treatment. Am J Otol 1987 May;8(3):201-202.
- 40. Sood S, Coles R. Hyperacusis and phonophobia in tinnitus patients. Br J Audiol 1998;22(1).
- 41. Khalfa S, Dubal S, Veuillet E, Perez-Diaz F, Jouvent R, Collet L. Psychometric normalization of a hyperacusis questionnaire. ORL J Otorhinolaryngol Relat Spec 2002 Nov-Dec;64(6):436-442.
- 42. Spitzer RL, Kroenke K, Williams JB, Patient Health Questionnaire Primary Care Study Group. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. JAMA 1999;282(18):1737-1744.
- 43. Spitzer RL, Kroenke K, Williams JB, Löwe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med 2006;166(10):1092-1097.
- 44. Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess 1985 02/01; 2014/11;49(1):71-75.
- 45. Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, et al. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care 2008 Mar;46(3):266-274.
- 46. Ritter P, Lorig K, Laurent D, Matthews K. Internet versus mailed questionnaires: a randomized comparison. J Med Internet Res 2004 Sep 15;6(3):e29.
- 47. Thoren ES, Andersson G, Lunner T. The use of research questionnaires with hearing impaired adults: online vs. paper-and-pencil administration. BMC Ear Nose Throat Disord 2012 Oct 29;12:12-6815-12-12.

- 48. Campbell M, Fitzpatrick R, Haines A, Kinmonth AL, Sandercock P, Spiegelhalter D, et al. Framework for design and evaluation of complex interventions to improve health.(Education and Debate). Br Med J 2000;321(7262):694.
- 49. Moore G, Audrey S, Barker M, Bond L, Bonell C, Hardeman W, et al. Process evaluation of complex interventions. Complex Interventions in Health: An Overview of Research Methods, 2015: 222.
- 50. Glasgow, R.E., Vogt, T.M. and Boles, S.M. (1999) Evaluating the public health impact of health promotion interventions: the RE-AIM framework, Am J Public Health, 89, 9, 1322-1327.
- 51. Dzewaltowski DA, Glasgow RE, Klesges LM, Estabrooks PA, Brock E. RE-AIM: evidence-based standards and a Web resource to improve translation of research into practice. Annals of Behavioral Medicine 2004;28(2):75-80.
- 52. Linnan L, Steckler AB. Process evaluation for public health interventions and research. Jossey-Bass San Francisco, CA; 2002.
- 53. Baranowski T, Stables G. Process evaluations of the 5-a-day projects. Health Educ Behav 2000 Apr;27(2):157-166.
- 54. Schulz KF, Altman DG, Moher D. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMC medicine 2010;8: 18-18.
- 55. Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. *Nurse education today* 2004; *24*(2), 105-112.
- 56. Teddlie C. Foundations of mixed methods research: Integrating quantitative and qualitative approaches in the social and behavioral sciences. Foundations of mixed methods research: 2009.
- 57. Office for National Statistics. Internet access: households and individuals. 2015; London: Her Majesty's Stationary Office.
- 58. Brown J, Michie S, Geraghty AW, Yardley L, Gardner B, Shahab L, et al. Internet-based intervention for smoking cessation (StopAdvisor) in people with low and high socioeconomic status: a randomised controlled trial. The Lancet Respiratory Medicine 2014;2(12):997-1006.
- 59. Moss-Morris R, McCrone P, Yardley L, van Kessel K, Wills G, Dennison L. A pilot randomised controlled trial of an Internet-based cognitive behavioural therapy self-management programme (MS Invigor8) for multiple sclerosis fatigue. Behav Res Ther 2012;50(6):415-421.